CLINICAL TRIAL: NCT00199134
Title: FRAGRANCE Trial(Femara Reanalysed Through Genomics for Response Assessment, Calibration and Empowerment)
Brief Title: FRAGRANCE Part A Safety: Study to Find a Genetic Signature of de Novo Resistance to Letrozole
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Collaborators: Feculdade de Medicina da Universidade de Sao Paulo - Brasil (Other); Hospital de Clinicas de Porto Alegre (Other); Hospital do Cancer, Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRAGRANCE; NCT00199199 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer
Keywords: neoadjuvant treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Letrozole (Other): Letrozole 2.5 mg per day
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Size of the tumor is followed

SUMMARY:
Find a genetic signature of de novo resistance to letrozole in adjuvant breast cancer;

DETAILED DESCRIPTION:
The aromatase inhibitors are drugs already approved for the treatment of breast cancer in the adjuvant and metastatic setting, and have demonstrated a superiority when compared to other hormone therapy agents as tamoxifen. FRAGRANCE is a trial of neoadjuvant hormone therapy activated in September 2004 at the Jules Bordet Institute. The main objective of this study is to find a genetic signature of de novo resistance to letrozole The standard dose of letrozol, 2,5 mg/day, is given orally during 4 months previous to the definitive breast surgery. The advantages of the neoadjuvant setting are a) the possibility to directly evaluate the response to therapy, which is of great value to decide adjuvant treatment; b) the increase chance of performing breast conserving surgery; c) and, because a tumor sample is obtained before and after treatment, the identification of predictive markers of response or resistance to treatment, including a genetic signature, obtained using the microarray technology. Eligible patients are women with early hormonal receptor positive breast cancer, with any contra-indication or refusal to the administration of chemotherapy The side effects of letrozole are already well known, and include more commonly hot flashes, nausea and vomiting, headache, arthralgia/myalgia, fatigue, and oedema. After surgery, adjuvant treatment will be done according to the standard practice of the Institute, considering the possibility of continuing letrozole for a total of at least 5 years, if a satisfactory response is achieved The first part of this trial will include 49 patients.

This trial will soon become a multicenter, multinational trial of 160 patients.

ELIGIBILITY:
Inclusion criteria :

1. Female gender
2. Post-menopausal(no age limit) defined as:

   1. Radiation-induced menopause or surgical bilateral oophorectomy, or
   2. Women with an intact uterus and

   i. > 55 years of age or ii. without menses for the last 5 years or iii. £ 55 years of age and has not had menses for at least the last 12 months (but has had menses in the last 5 years) and has postmenopausal levels of FSH c. Women without an intact uterus and i. > 55 years of age or ii. £ 55 years of age and has postmenopausal levels of FSH
3. Contraindications for the use of neoadjuvant/adjuvant chemotherapy, refusal by the patient to receive chemotherapy or if the investigator believes the patient is a suitable candidate for this protocol.
4. WHO performance status < 1
5. Histologically-confirmed ductal or lobular operable adenocarcinoma of the breast (stage I, II and III)
6. Confirmed absence of liver, lung and bone metastases.
7. Primary tumor of at least 2 cm, measured clinically and/or radiologically
8. Multifocal invasive tumors are not eligible, unless a biopsy showing ER positivity can be obtained from each tumor lesion.
9. ER-positive and/or PgR-positive tumors, defined according to immunohistochemistry (i.e. > 10% of positive cells after immunostaining), if woman younger 70 years; ER-positive or PgR-positive tumors if woman older than 70 years.
10. Fixed and frozen samples from the primary tumor, obtained before treatment, must be available for evaluation of biological markers (cDNA microarrays, EGFR, HER-2, intra-tumoral aromatase).
11. No concurrent second malignancy, including contralateral breast cancer (exceptions are: adequately treated basal cell carcinoma of the skin and in situ carcinoma of the cervix). Any prior second malignancy must be in remission for ³ 5 years.
12. No other serious illness or medical condition including:

    * History of documented congestive heart failure; angina pectoris requiring antianginal medication; evidence of recent (< 6 months) transmural infarction on ECG; poorly controlled hypertension (e.g. systolic >180 mm Hg or diastolic greater than 100 mm Hg); clinically significant valvular heart disease; or high-risk uncontrolled arrhythmias.
    * Chronic lung disease
    * History of significant neurological or psychiatric disorders that would prohibit the understanding and giving of informed consent, including psychotic disorders, mental retardation, and dementia.
    * Active concurrent infection
13. No concurrent or previous anti-cancer treatment is allowed
14. Adequate organ function as defined by:

    * Neutrophils ³ 1.5 x 109/L
    * Platelets ³ 100 x 109/L
    * Bilirubin £ 1.5x upper limit of normal (ULN)
    * Transaminases £ 2.5x ULN
    * Creatinine £ 1.5x ULN
15. Normal left ventricular ejection fraction by echocardiography or MUGA scan [for combination studies only]
16. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
17. Before patient registration/randomization, informed consent must be given according to ICH/EU GCP, and national/local regulations.

Exclusion crieria :

Non specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2004-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Response Rate Pathologic complete response rate | at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Christos Sotiriou, MD, PhD, Study Chair — Jules Bordet Institute
Locations (1):
- Jules Bordet Institute, Brussels, Belgium